CLINICAL TRIAL: NCT04532840
Title: Effect of Cryotherpy on Hypertrophic Scar
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zakria Mowafy (Other)
Responsible Party: Sponsor-Investigator, Zakria Mowafy, Professor of Physical Therapy for Surgery Faculty of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.t.REC/012/002266
Record Dates: First submitted 2020-08-18; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Hypertrophic Scars
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Cryotherapy; Patient Positioning; Massage

STUDY DESIGN:
Intervention Model Description: This study will be delimited in the following aspects:
  1. Subjects:
     Sixty patients suffering from hypertrophic scar will be randomly divided into two equal groups each one has 30 patients.
  2. Equipment and tools:
  2.1. Measurement equipment: Vancouver scar scale. MAPS (Matching Assessment of Scars and Photographs) (Masters et al., 2006). 2.2. Therapeutic equipment: Gymna Cryoflow ICE-CT. Temperature resistant polymide tape (48 wide)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (control group) (Active Comparator): This group includes 30 patients will receive routine medical treatment and routine physical therapy as (Exercising, Positioning and splinting, Pressure Therapy and Massage).
  Interventions: Other: Exercising, Positioning and splinting, Pressure Therapy and Massage
- Group B: (Study group) (Experimental): This group includes 30 patients will receive cryotherapy (at least 10 minutes at -14 degree , 2 sessions per week , for 10 weeks ) in addition to routine medical and physical therapy treatment.
  Interventions: Device: cryotherapy (Gymna Cryoflow ICE-CT); Other: Exercising, Positioning and splinting, Pressure Therapy and Massage

INTERVENTIONS:
Device: cryotherapy (Gymna Cryoflow ICE-CT) — Cryotherapy (also called cryoablation) method was produced by James Arnot in England in 1945 to reduce the size of cancerous cells based on the theory that cold blood cells destroy the cells. Campbell White of New York City used cryotherapy as the first dermatological indication in early-stage epithelioma patients in 1890. Later in 1907, Whitehouse described the use of this method in diferent diseases such as pigmented nevus and lupus. In addition, he has published a case series of skin cancers in different face regions.
  Other Names: Gymna Cryoflow ICE-CT
  Arms: Group B: (Study group)
Other: Exercising, Positioning and splinting, Pressure Therapy and Massage — Exercising, Positioning and splinting, Pressure Therapy and Massage

SUMMARY:
Purpose of the study:

The purpose of the study is to evaluate the therapeutic effect of cryotherpy in treating hypertrophic scar.

It will be hypothesized that:

Cryotherapy may not have an effect on hypertrophic scar.

DETAILED DESCRIPTION:
The potential of cryotherapy application in vitro data indicated that using freezing treatment on VFFs + TGF-β1 (myofibroblast) modulated ECM turnover toward antifibrosis and normalization, attenuated myofibroblast differentiation, reduced cell migration, and weakened the contractile activity. On both VFFs ± TGF-β1, freezing treatment raised LP regeneration (HAS1, decorin).

The findings indicate that cryotherapy may play a protective role in scar formation and contribute to lamina regeneration.

Furthermore the need of this study was developed from the lack in the quantitative knowledge and information in the published studies about the effect of cryotherapy on hypertrophic scar.

This study will be designed to provide a guideline about the effect of effect of cryotherapy on hypertrophic scar height, thickness and discoloration, and to assist in planning an ideal treatment regimen for reducing hypertrophic scar.

Delimitations:

This study will be delimited in the following aspects:

1. Subjects:

   Sixty patients suffering from hypertrophic scar will be randomly divided into two equal groups each one has 30 patients.
2. Equipment and tools:

2.1. Measurement equipment: Vancouver scar scale. MAPS (Matching Assessment of Scars and Photographs). 2.2. Therapeutic equipment: Gymna Cryoflow ICE-CT. Temperature resistant polymide tape (48 wide).

Hypothesis:

It will be hypothesized that:

Cryotherapy may not have an effect on hypertrophic scar.

Basic Assumptions:

It will be assumed that:

* All patients will receive the same kinds of medication and the same nursing care.
* All subjects are free from any chronic disease.
* All subjects will continue in the study.
* All patients will follow the instructions during the treatment

ELIGIBILITY:
Inclusion Criteria:

* Age range between 20- 40 years.
* Both sexes will participate in the study.
* All patients participated will begin treatment program one month after injury depending on injury characteristics.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* Diabetes mellitus.
* Individuals with cardiopulmonary conditions.
* Individuals undergoing radiation therapy or chemotherapy.
* Hepatic or pancreatic diseases.
* Sensory impairment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-09-15 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
scar height | 3 months
  The potential of cryotherapy application in vitro data indicated that using freezing treatment on scar decrease its height

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arno AI, Gauglitz GG, Barret JP, Jeschke MG. Up-to-date approach to manage keloids and hypertrophic scars: a useful guide. Burns. 2014 Nov;40(7):1255-66. doi: 10.1016/j.burns.2014.02.011. Epub 2014 Apr 24. PMID 24767715
- [Background] Atiyeh BS, Hayek SN, Gunn SW. New technologies for burn wound closure and healing--review of the literature. Burns. 2005 Dec;31(8):944-56. doi: 10.1016/j.burns.2005.08.023. Epub 2005 Nov 4. PMID 16274932